CLINICAL TRIAL: NCT06795542
Title: Predictive Factors for the Success of Transforaminal Epidural Injection in Lumbosacral Radiculopathy
Brief Title: The Aim of Study is to Identify the Predictive Factors for the Success of Transforaminal Epidural Injection in Treatment of Patients with Lumbosacral Radiculopathy
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Amr Mohamed Sedik (Other)
Responsible Party: Sponsor-Investigator, Amr Mohamed Sedik, Amr Mohamed Sedek Ahmed, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-1-05MS
Record Dates: First submitted 2025-01-18; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Radiculopathy
Keywords: predictive factors; transforaminal; epidural; injection
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: steroid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- lumbosacral transforaminal epidural injection (Experimental): Transforaminal Epidural Injections using C-arm imaging with or without Fluoroscopic Guidance
  Interventions: Procedure: lumbosacral transforaminal epidural injection at the level of L4-5, L5-S1, or S1 neural foramina

INTERVENTIONS:
Procedure: lumbosacral transforaminal epidural injection at the level of L4-5, L5-S1, or S1 neural foramina — The most widely used injection therapy is epidural injection of steroids, by either the interlaminar route or the caudal route. More contentious are transforaminal injections of steroids. These involve the injection of steroids directly and accurately onto the affected spinal nerve, under radiologic guidance. Meanwhile, transforaminal injection of steroids has been shown to be more effective than interlaminar injection of steroids

SUMMARY:
the aim of the study is to identify predictive factors for the success of transforaminal epidural injection in the treatment of patients with lumbosacral radiculopathy

DETAILED DESCRIPTION:
Lumbar radicular pain (known as sciatica) represents a prevalent medical and socioeconomic problem.

More than half of the patients with sciatica report a decline in their activities of daily living and ability to work.

Mixed Pathologies as foraminal stenosis, spondylolisthesis, and space-occupying lesions in the lumbar spine can cause Sciatica but the most common cause is lumbar disc herniation. (1) Overall, the vast majority of patients with lumbosacral radiculopathy recover with conservative care as trial of bed rest, oral medications, lumbar corsets and physiotherapy. (2) The involvement of inflammation has attracted the use of steroids (corticosteroids) to reduce the inflammation and, thereby, relieve the pain. Injections of steroids, by various routes, have been used as an alternative to surgery, and as an alternative or complement to conservative therapy, for the treatment of lumbar radicular pain. (3) Steroids are believed to have a therapeutic effect due to their anti inflammatory properties.

This belief is supported by evidence from in vitro studies that show that steroids have a role in decreasing inflammatory mediators such as cytokines and chemokines another study suggests that steroids may provide a stabilizing effect on nociceptive signaling in C-fibers and suppression of ectopic neural discharges. (4) The most widely used injection therapy is epidural injection of steroids, by either the interlaminar route or the caudal route. More contentious are transforaminal injections of steroids. These involve the injection of steroids directly and accurately onto the affected spinal nerve, under radiologic guidance. Meanwhile, transforaminal injection of steroids has been shown to be more effective than interlaminar injection of steroids (5) Transforaminal epidural injection may be by autologous Platelet Rich Plasma (PRP) as a novel pharmaceutical agent that has strongly emerged in recent years to treat patients of lumbar disc herniation.(6)

ELIGIBILITY:
Inclusion Criteria:

- 1.Patients who underwent lumbosacral transforaminal epidural injection at the level of L4-5, L5-S1, or S1 neural foramina 2.Patients age 18 to 60 years 3.Patients had been symptomatic longer than 6 Weeks with Leg pain more than back pain with failure conservative treatment.

4.Patients had undergone an MRI Lumbosacral imaging scan documenting disc prolapse

Exclusion Criteria:

* 1- Patients had previous lumbar surgery 2- Patients had a large herniated disc with severe central or foraminal stenosis on magnetic resonance imaging 3- Patients had Scoliosis , spondylolisthesis or malignancy 4- patients with neurological deficit. 5-Patients had a blood coagulation disorder, or had experienced an allergic reaction to local anesthetics or corticosteroids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Transformainal Epidural Injection | 3 months
  All patients will be followed up in outpatient clinic every 2 weeks for 3months by assessing Visual Analogue Pain Scale (VAS)
Transformainal Epidural Injection | 3 months
  All patients will be followed up in outpatient clinic every 2 weeks for 3months by assessing
  -Roland & Morris Disability Questionnaire
Transformainal Epidural Injection | 3 months
  All patients will be followed up in outpatient clinic every 2 weeks for 3months by assessing modified oswestry disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Neurossurgery Department of Sohag university, Sohag, Sohag Governorate, Egypt